CLINICAL TRIAL: NCT05155865
Title: Conduction System Pacing Versus Biventricular Pacing for Cardiac ResYNChronization (CSP-SYNC)
Brief Title: Conduction System Pacing Versus Biventricular Pacing for Cardiac ResYNChronization
Acronym: CSP-SYNC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, David Žižek, MD, PhD, assist. prof. David Žižek, MD, PhD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSP-SYNC
Record Dates: First submitted 2021-11-30; First posted 2021-12-14 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Dilated Cardiomyopathy with Conduction Defect; Left Bundle-Branch Block; Heart Failure; Resynchronization Therapy; Cardiac Remodeling, Ventricular
Keywords: left bundle branch block; dilated cardiomyopathy; resynchronization therapy; myocardial work; arrhythmia
MeSH Terms: conditions — Idiopathic dilation cardiomyopathy; Bundle-Branch Block; Heart Failure; Ventricular Remodeling; Cardiomyopathy, Dilated; Arrhythmias, Cardiac | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Resynchronization with conduction system pacing (Experimental): Implantation of permanent pacemaker with conduction system pacing (preferably left bundle branch) with or without defibrillator lead placement. Optimal guidelines-based heart failure treatment and antiarrhythmic drugs.
  Interventions: Device: Resynchronization with conduction system pacing
- Cardiac resynchronization therapy with biventricular stimulation (Active Comparator): Implantation of cardiac resynchronization therapy with biventricular stimulation with or without defibrillator lead placement. Optimal guidelines-based heart failure treatment and antiarrhythmic drugs.
  Interventions: Device: Cardiac resynchronization therapy with biventricular stimulation

INTERVENTIONS:
Device: Resynchronization with conduction system pacing — Implantation of permanent pacemaker with conduction system pacing (preferably left bundle branch) with or without defibrillator lead placement
  Arms: Resynchronization with conduction system pacing
Device: Cardiac resynchronization therapy with biventricular stimulation — Implantation of cardiac resynchronization therapy with biventricular stimulation with or without defibrillator lead placement
  Arms: Cardiac resynchronization therapy with biventricular stimulation

SUMMARY:
Cardiac resynchronization therapy (CRT) with biventricular pacing (BiV) is the cornerstone treatment for heart failure patients with ventricular dyssynchrony. Recently, a new concept, conduction system pacing (CSP) with permanent pacing, including His bundle pacing and left bundle branch pacing, has been proposed as a potential alternative to conventional BiV-CRT. The prospective, randomized trial will compare echocardiographic, electrocardiographic, and clinical effects of CSP versus conventional BiV pacing in heart failure patients with reduced ejection fraction (LVEF ≤ 35%), sinus rhythm, and left bundle branch block. Patients will be randomized to either CSP or biventricular pacing study group and followed up for at least 6 months. The study will explore whether CSP is non-inferior to BiV pacing in echocardiographic, electrocardiographic, and clinical outcomes.

DETAILED DESCRIPTION:
Cardiac resynchronization therapy (CRT) with biventricular pacing is an integral part of heart failure therapy in patients with reduced ejection fraction and wide QRS. Previous studies have demonstrated improved quality of life, reduced heart failure hospitalization, and decreased all-cause mortality. However, approx. 30% of patients still do not benefit from this therapy. High pacing thresholds and phrenic nerve stimulation are also common problems with BiV stimulation. Newer CRT systems with improved programmability and algorithms in conjunction with quadripolar left ventricular leads have solved some challenges of BiV pacing. However, BiV stimulation with non-physiological epicardial activation has shown a possible pro-arrhythmic effect which is more pronounced in the non-responder population.

On the other hand, CSP provides synchronous physiological ventricular activation with possible superior electrical and mechanical resynchronization compared to BiV pacing. Electrical activation maps obtained during CSP showed normalization of left bundle branch block with more homogeneous electrical resynchronization than in biventricular pacing. Additionally, BiV CRT effectively corrects mechanical dyssnchrony, demonstrated with homogenization of myocardial work. This has already been proven as the underlying pathophysiological mechanism for successful CRT response. However, the effect of CSP on echocardiographic parameters of mechanical dyssynchrony is not known.

Previous studies of CSP focused on feasibility and its benefits over right ventricular pacing in patients with refractory atrial fibrillation who underwent atrioventricular node ablation and pacemaker implantation. Promising results were followed by the acknowledgment of this physiological mode of pacing by the recent guidelines of European Society of Cardiology. However, studies evaluating the value of CSP as an alternative approach to BiV CRT in heart failure patients are limited. The purpose of this study is to compare the effects of CSP and conventional BiV pacing on electrocardiographic and echocardiographic parameters as well as on clinical outcomes in patients with heart failure with reduced ejection fraction (LVEF ≤35%), sinus rhythm, and left bundle branch block. In this single-center study, 60 patients will be randomized into one of two arms: a BiV pacing arm with BiV CRT implantation based on clinical guidelines or an experimental CSP arm with the implantation of a CSP device. Device with a defibrillator (ICD) will be selected at the discretion of the implanting physician. Baseline and follow up assessments will include clinical evaluation (New York Heart Association class, 6-minute walking distance), evaluation of quality of life (EQ-5D index), laboratory tests (N-terminal pro-B-type natriuretic peptide), electrocardiographic recordings (standard 12-leads ECG and high-resolution-ECG), and echocardiographic evaluation (standard echocardiographic parameters of LV reverse remodeling and non-invasive myocardial work assessment). Intra-operative and procedural parameters will also be recorded.

Investigators hypothesize that CSP could represent a feasible and safe alternative to conventional BiV pacing in terms of clinical, electrocardiographic, and echocardiographic outcomes.

ELIGIBILITY:
Inclusion Criteria:

The proposed inclusion criteria represent the minimum recommendations for CRT implantation according to the ESC 2021 guidelines. In addition:

1. Sinus rhythm and complete left bundle branch block according to Strauss criteria
2. LVEF ≤35%
3. NYHA class II-III
4. Optimal medical heart failure therapy for at least 3 months before enrollment
5. The patient is able to understand and willing to provide a written informed consent
6. 18 years of age or older

Exclusion Criteria:

1. Mechanical tricuspid valve replacement
2. More than moderate valvular disease
3. Unstable angina, acute MI, CABG, or PCI within the past 6 months
4. Persistent or permanent atrial fibrillation
5. Ventricular arrhythmias (frequent PVC) which do not allow to acquire consecutive regular beats during echocardiography and electrocardiography
6. Higher degree AV block
7. Life expectancy of less than 12 months
8. Pregnancy and breastfeeding
9. Acute illness or active systemic infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Change in left ventricular volume | acute after the procedure, 1 month, 6 months, 12 months
  Effect on reverse left ventricular remodeling measured as changes in left ventricular volume in both arms
Change in left ventricular ejection fraction | acute procedure, 1 month, 6 months, 12 months
  Effect on reverse left ventricular remodeling measured as changes in left ventricular ejection fraction in both arms
Difference in Heart Failure Class | 6 months
  From class 1 to 4
Difference in pro-BNP value | 6 months
  pg/mL
Difference in 6-minute walk test distance | 6 months
  meters
Difference in the EQ-5D index | 6 months
  score

SECONDARY OUTCOMES:
Difference in myocardial work redistribution | acute after the procedure, 1 month, 6 months, 12 months
  Echo measurement
Difference in QRS complex width | acute after the procedure, 1 month, 6 months, 12 months
  ms
Difference in filtered QRS duration on high-resolution electrocardiogram | acute after procedure, 1 month, 6 months, 12 months
  ms
Difference in sum absolute QRST integral | acute after the procedure, 1 month, 6 months, 12 months
  ms
Difference in arrhythmia occurrence | at least 12 months after enrollment
  Descriptive
Rate of procedural complications | at least 12 months after enrollment
  Descriptive
Tpeak-end duration | acute after the procedure, 1 month, 6 months, 12 months
  ms

CONTACTS AND LOCATIONS:
Overall Officials: Marta Cvijc, MD, Study Chair — University Medical Centre Ljubljana (Slovenia); Anja Zupan Meznar, MD, Study Chair — University Medical Centre Ljubljana (Slovenia)
Locations (1):
- University medical centre Ljubljana, Ljubljana, Slovenia, Slovenia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Sharma PS, Vijayaraman P. Conduction System Pacing for Cardiac Resynchronisation. Arrhythm Electrophysiol Rev. 2021 Apr;10(1):51-58. doi: 10.15420/aer.2020.45. PMID 33936744
- [Background] Herweg B, Welter-Frost A, Vijayaraman P. The evolution of cardiac resynchronization therapy and an introduction to conduction system pacing: a conceptual review. Europace. 2021 Apr 6;23(4):496-510. doi: 10.1093/europace/euaa264. PMID 33247913
- [Background] Wu S, Su L, Vijayaraman P, Zheng R, Cai M, Xu L, Shi R, Huang Z, Whinnett ZI, Huang W. Left Bundle Branch Pacing for Cardiac Resynchronization Therapy: Nonrandomized On-Treatment Comparison With His Bundle Pacing and Biventricular Pacing. Can J Cardiol. 2021 Feb;37(2):319-328. doi: 10.1016/j.cjca.2020.04.037. Epub 2020 May 7. PMID 32387225
- [Background] Vinther M, Risum N, Svendsen JH, Mogelvang R, Philbert BT. A Randomized Trial of His Pacing Versus Biventricular Pacing in Symptomatic HF Patients With Left Bundle Branch Block (His-Alternative). JACC Clin Electrophysiol. 2021 Nov;7(11):1422-1432. doi: 10.1016/j.jacep.2021.04.003. Epub 2021 Apr 25. PMID 34167929
- [Background] Deif B, Ballantyne B, Almehmadi F, Mikhail M, McIntyre WF, Manlucu J, Yee R, Sapp JL, Roberts JD, Healey JS, Leong-Sit P, Tang AS. Cardiac resynchronization is pro-arrhythmic in the absence of reverse ventricular remodelling: a systematic review and meta-analysis. Cardiovasc Res. 2018 Sep 1;114(11):1435-1444. doi: 10.1093/cvr/cvy182. PMID 30010807
- [Background] Galand V, Singh JP, Leclercq C. Alternative left ventricular pacing approaches for optimal cardiac resynchronization therapy. Heart Rhythm. 2019 Aug;16(8):1281-1289. doi: 10.1016/j.hrthm.2019.03.011. Epub 2019 Mar 16. PMID 30885737
- [Background] Duchenne J, Aalen JM, Cvijic M, Larsen CK, Galli E, Bezy S, Beela AS, Unlu S, Pagourelias ED, Winter S, Hopp E, Kongsgard E, Donal E, Fehske W, Smiseth OA, Voigt JU. Acute redistribution of regional left ventricular work by cardiac resynchronization therapy determines long-term remodelling. Eur Heart J Cardiovasc Imaging. 2020 Jun 1;21(6):619-628. doi: 10.1093/ehjci/jeaa003. PMID 32031587
- [Background] Cvijic M, Duchenne J, Unlu S, Michalski B, Aarones M, Winter S, Aakhus S, Fehske W, Stankovic I, Voigt JU. Timing of myocardial shortening determines left ventricular regional myocardial work and regional remodelling in hearts with conduction delays. Eur Heart J Cardiovasc Imaging. 2018 Aug 1;19(8):941-949. doi: 10.1093/ehjci/jex325. PMID 29272366
- [Background] Abdelrahman M, Subzposh FA, Beer D, Durr B, Naperkowski A, Sun H, Oren JW, Dandamudi G, Vijayaraman P. Clinical Outcomes of His Bundle Pacing Compared to Right Ventricular Pacing. J Am Coll Cardiol. 2018 May 22;71(20):2319-2330. doi: 10.1016/j.jacc.2018.02.048. Epub 2018 Mar 10. PMID 29535066
- [Background] Dandamudi G, Vijayaraman P. History of His bundle pacing. J Electrocardiol. 2017 Jan-Feb;50(1):156-160. doi: 10.1016/j.jelectrocard.2016.09.011. Epub 2016 Sep 24. PMID 27720211
- [Background] Brugada J, Katritsis DG, Arbelo E, Arribas F, Bax JJ, Blomstrom-Lundqvist C, Calkins H, Corrado D, Deftereos SG, Diller GP, Gomez-Doblas JJ, Gorenek B, Grace A, Ho SY, Kaski JC, Kuck KH, Lambiase PD, Sacher F, Sarquella-Brugada G, Suwalski P, Zaza A; ESC Scientific Document Group. 2019 ESC Guidelines for the management of patients with supraventricular tachycardiaThe Task Force for the management of patients with supraventricular tachycardia of the European Society of Cardiology (ESC). Eur Heart J. 2020 Feb 1;41(5):655-720. doi: 10.1093/eurheartj/ehz467. No abstract available. PMID 31504425